CLINICAL TRIAL: NCT04702945
Title: Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN) - Population-based Registry of Suspected and Confirmed COVID-19 Cases
Brief Title: Canadian COVID-19 Emergency Department Registry
Acronym: CCEDRRN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Genome British Columbia (Industry); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other)
Responsible Party: Principal Investigator, Corinne Hohl, Associate Professor, University of British Columbia
Other Study IDs: H20-01015
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Covid-19
Keywords: Coronavirus; Infectious diseases; Registry
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry participants: Patients presenting to participating emergency departments with suspected and or confirmed COVID-19.

SUMMARY:
Coronavirus Disease 2019 (COVID -19) is the largest public health crisis in over a century. There is an urgent need for high-quality population-level data to understand modifiable risks for disease severity, transmissibility, and to develop evidence-based prevention (i.e. vaccination), treatment and resource allocation strategies.

The Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN) created a population-based registry of suspected and confirmed consecutive cases of COVID-19. The purpose of this registry is to derive and validate clinical decision rules, evaluate diagnostic tests and vaccine effectiveness, and complete cohort, case-control and observational studies to inform the pandemic response.

DETAILED DESCRIPTION:
This national multi-centre registry is designed to enroll population-based consecutive eligible patients presenting with suspected or confirmed COVID-19 to 50 emergency departments in eight Canadian provinces from March 1 2020 and data collection is ongoing for the duration of the pandemic.

Data will be abstracted from the medical chart and entered into a central, web-based REDCap database. The investigators adopted the ISARIC variables into the database where there was a match. The investigators will develop standardized operating procedures for screening of potentially eligible patients, data entry and follow-up. Current data dictionaries are kept on the registry's website (https://canadiancovid19registry.org/).

At 30 days, the investigators will contact patients by telephone to obtain verbal consent for follow-up. The investigators will measure the Veterans Rand 12-item Health Survey (VR12), calculate the WHO Ordinal Outcome Scale and ask contextual questions in consenting patients. The VR12 will be measured at 60 days, and 6 and 12 months. The contextual questions were developed with input from patients with lived experience with COVID-19 infection and addressed cultural, racial, gender, socioeconomic and self-isolation issues.

The Health Data Research Network facilitated the development of a unique data flow of personal health identifiers and study identification numbers from each province for all participating institutes. This will allow linkage of registry data with national administrative data repositories.

ELIGIBILITY:
The investigators defined two periods for enrollment based on the availability of COVID-19 testing. Research assistants used medical microbiology testing and discharge diagnoses to screen for potentially eligible patients.

In Period 1, COVID-19 testing in each province was restricted to specific patient populations (e.g., healthcare workers, admitted patients).

Inclusion Criteria:

* Meeting the WHO suspect COVID-19 criteria: Fever (self-reported or subjective fever) and at least one symptom/sign of respiratory illness (e.g., flu-like illness, cough, shortness of breath)
* Presenting to the emergency department and tested for COVID-19 in the emergency department

No exclusion criteria in Period 1

Period 2 started on the date which each province expanded testing criteria allowing clinicians to test patients based on clinical suspicion or policy.

Inclusion Criteria:

* Presenting to the emergency department within 14 days of a positive COVID-19 (by self-report or in medical chart) and presents with clinical symptoms consistent with COVID-19
* Tested for COVID-19 in the emergency department, or within 24 hours after emergency department arrival.

Exclusion Criteria

* Patients tested for COVID-19 in the context of an elective admission (e.g., planned hip revision)
* Patients tested for COVID-19 and seen in the emergency department directly by another service (e.g., trauma team activation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to participating Canadian emergency departments with suspected and or confirmed COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed COVID-19 diagnosis | 14 days
  Biological specimen is tested positive for SARS-CoV-2 using reverse transcription polymerase chain reaction (RT PCR). The specimen had to be drawn within two weeks of the emergency department visit if the patient presented with a COVID-19-related complication. If the initial test was negative, the patient had to have a positive specimen within 14 days of the index visit.

SECONDARY OUTCOMES:
Hospital admission | 30 days
  Any hospital admission within 30 days of index emergency department visit captured in medical chart.
Mechanical ventilation | 30 days
  Any mechanical ventilation during any hospital visit within 30 days of index emergency department visit captured in medical chart.
Emergency department revisits | 30 days
  Any emergency department revisits within 30 days of index emergency department visit captured in medical chart.
Hospital re-admissions | 30 days
  Any hospital re-admissions within 30 days of index emergency department visit date captured in medical chart.
30 day mortality | 30 days
  Any death captured within 30 days of index emergency department visit captured by medical charts.
Clinical recovery | 30 days
  Captured through telephone follow-up using the World Health Organization Ordinal Outcome Scale at 30 days after index emergency department visit. The scale is scored from 1 to 8 ('1'= no limitations to activities, '8'=death) to measure clinical improvement at 30 days.
Patient quality of life | 12 months
  Captured through telephone follow-up using the Veterans Rand 12-item Health Survey at 30 days, 60 days, and 6 and 12 months after index emergency department visit.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne M Hohl, MD, MSc, Principal Investigator — University of British Columbia
Locations (50):
- Canada (50):
  - Foothills Medical Centre, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Northeast Community Health Centre, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Abbotsford Regional Hospital, Abbotsford, British Columbia
  - Royal Inland Hospital, Kamloops, British Columbia
  - Kelowna General Hospital, Kelowna, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Eagle Ridge Hospital, Port Moody, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Mount Saint Joseph Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dartmouth General Hospital, Dartmouth, Nova Scotia
  - Halifax Infirmary, Halifax, Nova Scotia
  - Cobequid Community Health Centre, Lower Sackville, Nova Scotia
  - Hants Community Hospital, Windsor, Nova Scotia
  - Health Science North, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre (University Hospital), London, Ontario
  - London Health Sciences Centre (Victoria Hospital), London, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - Hôpital du Sacré-Coeur, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Montréal General Hospital (MUHC), Montreal, Quebec
  - Royal Victoria Hospital (MUHC), Montreal, Quebec
  - Centre Hospitalier de l'Université Laval (CHU de Québec), Québec, Quebec
  - Hôpital de l'Enfant-Jésus (CHU de Québec), Québec, Quebec
  - Hôpital du Saint-Sacrement (CHU de Québec), Québec, Quebec
  - Hôpital Saint-François d'Assise (CHU de Québec), Québec, Quebec
  - Hôtel-Dieu de Québec (CHU de Québec), Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - Pasqua Hospital, Regina, Saskatchewan
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University, Saskatoon, Saskatchewan
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
  - St Paul's Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Rosychuk RJ, Khangura JK, Ortiz SS, Cheng I, Bielska IA, Yan J, Morrison LJ, Hayward J, Grant L, Hohl CM; Canadian COVID-19 Rapid Response Network (CCEDRRN) for the Network of Canadian Emergency Researchers (NCER). Characteristics and outcomes of patients with COVID-19 who return to the emergency department: a multicentre observational study by the Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN). Emerg Med J. 2024 Mar 21;41(4):210-217. doi: 10.1136/emermed-2023-213277. PMID 38365437
- [Derived] Hohl CM, Cragg A, Purssell E, McAlister FA, Ting DK, Scheuermeyer F, Stachura M, Grant L, Taylor J, Kanu J, Hau JP, Cheng I, Atzema CL, Bola R, Morrison LJ, Landes M, Perry JJ, Rosychuk RJ; Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN) investigators for the Network of Canadian Emergency Researchers; Canadian Critical Care Trials Group. Comparing methods to classify admitted patients with SARS-CoV-2 as admitted for COVID-19 versus with incidental SARS-CoV-2: A cohort study. PLoS One. 2023 Sep 26;18(9):e0291580. doi: 10.1371/journal.pone.0291580. eCollection 2023. PMID 37751455
- [Derived] Archambault PM, Rosychuk RJ, Audet M, Bola R, Vatanpour S, Brooks SC, Daoust R, Clark G, Grant L, Vaillancourt S, Welsford M, Morrison LJ, Hohl CM; Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN) investigators; Network of Canadian Emergency Researchers; Canadian Critical Care Trials Group. Accuracy of Self-Reported COVID-19 Vaccination Status Compared With a Public Health Vaccination Registry in Quebec: Observational Diagnostic Study. JMIR Public Health Surveill. 2023 Jun 16;9:e44465. doi: 10.2196/44465. PMID 37327046
- [Derived] Lin K, Xu K, Daoust R, Taylor J, Rosychuk RJ, Hau JP, Davis P, Clark G, McRae AD, Hohl CM; Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN) investigators for the Network of Canadian Emergency Researchers, the Canadian Critical Care Trials Group. Prognostic association between d-dimer thresholds and 30-day pulmonary embolism diagnosis among emergency department patients with suspected SARS-CoV-2 infection: a Canadian COVID-19 Emergency Department Rapid Response Network study. CJEM. 2023 Feb;25(2):134-142. doi: 10.1007/s43678-022-00440-8. Epub 2023 Jan 10. PMID 36624252
- [Derived] Davis P, Rosychuk R, Hau JP, Cheng I, McRae AD, Daoust R, Lang E, Turner J, Khangura J, Fok PT, Stachura M, Brar B, Hohl CM; CCEDRRN investigators, and for the Network of Canadian Emergency Researchers and the Canadian Critical Care Trials Group. Diagnostic yield of screening for SARS-CoV-2 among patients admitted to hospital for alternate diagnoses: an observational cohort study. BMJ Open. 2022 Aug 10;12(8):e057852. doi: 10.1136/bmjopen-2021-057852. PMID 35948378
- [Derived] Hohl CM, Rosychuk RJ, Hau JP, Hayward J, Landes M, Yan JW, Ting DK, Welsford M, Archambault PM, Mercier E, Chandra K, Davis P, Vaillancourt S, Leeies M, Small S, Morrison LJ; Canadian COVID-19 Rapid Response Network (CCEDRRN) investigators for the Network of Canadian Emergency Researchers, for the Canadian Critical Care Trials Group. Treatments, resource utilization, and outcomes of COVID-19 patients presenting to emergency departments across pandemic waves: an observational study by the Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN). CJEM. 2022 Jun;24(4):397-407. doi: 10.1007/s43678-022-00275-3. Epub 2022 Apr 1. PMID 35362857
- [Derived] Hohl CM, Rosychuk RJ, Archambault PM, O'Sullivan F, Leeies M, Mercier E, Clark G, Innes GD, Brooks SC, Hayward J, Ho V, Jelic T, Welsford M, Sivilotti MLA, Morrison LJ, Perry JJ; Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN) investigators for the Network of Canadian Emergency Researchers and the Canadian Critical Care Trials Group. The CCEDRRN COVID-19 Mortality Score to predict death among nonpalliative patients with COVID-19 presenting to emergency departments: a derivation and validation study. CMAJ Open. 2022 Feb 8;10(1):E90-E99. doi: 10.9778/cmajo.20210243. Print 2022 Jan-Mar. PMID 35135824
- [Derived] McRae AD, Hohl CM, Rosychuk R, Vatanpour S, Ghaderi G, Archambault PM, Brooks SC, Cheng I, Davis P, Hayward J, Lang E, Ohle R, Rowe B, Welsford M, Yadav K, Morrison LJ, Perry J; Canadian COVID-19 Emergency Department Rapid Response Network (CCEDRRN) investigators for the Network of Canadian Emergency Researchers and the Canadian Critical Care Trials Group. CCEDRRN COVID-19 Infection Score (CCIS): development and validation in a Canadian cohort of a clinical risk score to predict SARS-CoV-2 infection in patients presenting to the emergency department with suspected COVID-19. BMJ Open. 2021 Dec 2;11(12):e055832. doi: 10.1136/bmjopen-2021-055832. PMID 34857584
- [Derived] Hohl CM, Rosychuk RJ, McRae AD, Brooks SC, Archambault P, Fok PT, Davis P, Jelic T, Turner JP, Rowe BH, Mercier E, Cheng I, Taylor J, Daoust R, Ohle R, Andolfatto G, Atzema C, Hayward J, Khangura JK, Landes M, Lang E, Martin I, Mohindra R, Ting DK, Vaillancourt S, Welsford M, Brar B, Dahn T, Wiemer H, Yadav K, Yan JW, Stachura M, McGavin C, Perry JJ, Morrison LJ; Canadian COVID-19 Emergency Department Rapid Response Network investigators and for the Network of Canadian Emergency Researchers and the Canadian Critical Care Trials Group. Development of the Canadian COVID-19 Emergency Department Rapid Response Network population-based registry: a methodology study. CMAJ Open. 2021 Mar 17;9(1):E261-E270. doi: 10.9778/cmajo.20200290. Print 2021 Jan-Mar. PMID 33731427